CLINICAL TRIAL: NCT04124471
Title: Positive Airway Pressure for the Treatment of the Obstructive Sleep Apnea Syndrome in Children With Down Syndrome (Stage 1)
Brief Title: Investigating the Experience of Living With Down Syndrome and Obstructive Sleep Apnea Syndrome (Stage 1)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Pennsylvania (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-016222; R61HL151253-01 (NIH)
Record Dates: First submitted 2019-10-04; First posted 2019-10-11 (Actual); Results first posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Down Syndrome; Obstructive Sleep Apnea
Keywords: Down Syndrome; Obstructive Sleep Apnea
MeSH Terms: conditions — Down Syndrome; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants treated with PAP (Other): This is a qualitative study for participants with Down Syndrome who use PAP to treat obstructive sleep apnea syndrome.
  Interventions: Behavioral: Open-ended semi-structured interviews

INTERVENTIONS:
Behavioral: Open-ended semi-structured interviews — Semi-structured interviews will explore such key constructs as knowledge/belief about OSAS and PAP therapy, routines and resources that promote or limit PAP use, barriers, self-efficacy, and communication and attitudes about PAP. The interviews will be performed with the parent and that they will be audio-recorded.

SUMMARY:
To identify the perceptions, beliefs, and family-relevant outcomes regarding the treatment of obstructive sleep apnea syndrome (OSAS) with positive airway pressure (PAP) in children with Down's Syndrome (DS).

DETAILED DESCRIPTION:
This is a multi-center outpatient study to be performed at two clinical sites: Children's Hospital of Philadelphia and Cincinnati Children's Hospital. Forty Caregivers of children with DS and OSAS treated with PAP and their children will be enrolled. The study comprises one 30-minute open-ended semi-structured interview per caregiver. The duration of the interview is approximate. It will last up to 30 minutes as some families may want to include more details.

ELIGIBILITY:
Inclusion Criteria -- Patients

* Children with DS and OSAS treated with PAP for at least 6 months
* Children aged between 6 and 17.5 years
* English proficiency

Inclusion Criteria -- Caregivers

* Parent or legal guardian of an eligible patient subject
* English proficiency
* Must live with the patient subject at least 4 nights of the week

Exclusion Criteria -- Patients

* In foster care
* Diagnosed with major illness, such as leukemia or severe cyanotic congenital heart disease listed for cardiac transplant as these severe diseases may add confounders

Exclusion Criteria -- Caregivers

* Foster parent

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Presson AP, Partyka G, Jensen KM, Devine OJ, Rasmussen SA, McCabe LL, McCabe ER. Current estimate of Down Syndrome population prevalence in the United States. J Pediatr. 2013 Oct;163(4):1163-8. doi: 10.1016/j.jpeds.2013.06.013. Epub 2013 Jul 23. PMID 23885965
- [Background] Mai CT, Kucik JE, Isenburg J, Feldkamp ML, Marengo LK, Bugenske EM, Thorpe PG, Jackson JM, Correa A, Rickard R, Alverson CJ, Kirby RS; National Birth Defects Prevention Network. Selected birth defects data from population-based birth defects surveillance programs in the United States, 2006 to 2010: featuring trisomy conditions. Birth Defects Res A Clin Mol Teratol. 2013 Nov;97(11):709-25. doi: 10.1002/bdra.23198. No abstract available. PMID 24265125
- [Background] de Graaf G, Buckley F, Skotko BG. Estimates of the live births, natural losses, and elective terminations with Down syndrome in the United States. Am J Med Genet A. 2015 Apr;167A(4):756-67. doi: 10.1002/ajmg.a.37001. PMID 25822844
- [Background] Sherman SL, Allen EG, Bean LH, Freeman SB. Epidemiology of Down syndrome. Ment Retard Dev Disabil Res Rev. 2007;13(3):221-7. doi: 10.1002/mrdd.20157. PMID 17910090
- [Background] Bull MJ; Committee on Genetics. Health supervision for children with Down syndrome. Pediatrics. 2011 Aug;128(2):393-406. doi: 10.1542/peds.2011-1605. Epub 2011 Jul 25. PMID 21788214
- [Background] Marcus CL, Carroll JL, Koerner CB, Hamer A, Lutz J, Loughlin GM. Determinants of growth in children with the obstructive sleep apnea syndrome. J Pediatr. 1994 Oct;125(4):556-62. doi: 10.1016/s0022-3476(94)70007-9. PMID 7931873
- [Background] Marcus CL, Greene MG, Carroll JL. Blood pressure in children with obstructive sleep apnea. Am J Respir Crit Care Med. 1998 Apr;157(4 Pt 1):1098-103. doi: 10.1164/ajrccm.157.4.9704080. PMID 9563725
- [Background] Amin RS, Kimball TR, Bean JA, Jeffries JL, Willging JP, Cotton RT, Witt SA, Glascock BJ, Daniels SR. Left ventricular hypertrophy and abnormal ventricular geometry in children and adolescents with obstructive sleep apnea. Am J Respir Crit Care Med. 2002 May 15;165(10):1395-9. doi: 10.1164/rccm.2105118. PMID 12016102
- [Background] Amin RS, Carroll JL, Jeffries JL, Grone C, Bean JA, Chini B, Bokulic R, Daniels SR. Twenty-four-hour ambulatory blood pressure in children with sleep-disordered breathing. Am J Respir Crit Care Med. 2004 Apr 15;169(8):950-6. doi: 10.1164/rccm.200309-1305OC. Epub 2004 Feb 5. PMID 14764433
- [Background] Miman MC, Kirazli T, Ozyurek R. Doppler echocardiography in adenotonsillar hypertrophy. Int J Pediatr Otorhinolaryngol. 2000 Aug 11;54(1):21-6. doi: 10.1016/s0165-5876(00)00338-4. PMID 10960692
- [Background] Tal A, Leiberman A, Margulis G, Sofer S. Ventricular dysfunction in children with obstructive sleep apnea: radionuclide assessment. Pediatr Pulmonol. 1988;4(3):139-43. doi: 10.1002/ppul.1950040304. PMID 2836784
- [Background] Gozal D, Kheirandish-Gozal L, Bhattacharjee R, Spruyt K. Neurocognitive and endothelial dysfunction in children with obstructive sleep apnea. Pediatrics. 2010 Nov;126(5):e1161-7. doi: 10.1542/peds.2010-0688. Epub 2010 Oct 18. PMID 20956420
- [Background] Kheirandish-Gozal L, Bhattacharjee R, Kim J, Clair HB, Gozal D. Endothelial progenitor cells and vascular dysfunction in children with obstructive sleep apnea. Am J Respir Crit Care Med. 2010 Jul 1;182(1):92-7. doi: 10.1164/rccm.200912-1845OC. Epub 2010 Mar 4. PMID 20203242
- [Background] Montgomery-Downs HE, Crabtree VM, Gozal D. Cognition, sleep and respiration in at-risk children treated for obstructive sleep apnoea. Eur Respir J. 2005 Feb;25(2):336-42. doi: 10.1183/09031936.05.00082904. PMID 15684300
- [Background] Chervin RD, Ruzicka DL, Giordani BJ, Weatherly RA, Dillon JE, Hodges EK, Marcus CL, Guire KE. Sleep-disordered breathing, behavior, and cognition in children before and after adenotonsillectomy. Pediatrics. 2006 Apr;117(4):e769-78. doi: 10.1542/peds.2005-1837. PMID 16585288
- [Background] Marcus CL, Radcliffe J, Konstantinopoulou S, Beck SE, Cornaglia MA, Traylor J, DiFeo N, Karamessinis LR, Gallagher PR, Meltzer LJ. Effects of positive airway pressure therapy on neurobehavioral outcomes in children with obstructive sleep apnea. Am J Respir Crit Care Med. 2012 May 1;185(9):998-1003. doi: 10.1164/rccm.201112-2167OC. Epub 2012 Feb 9. PMID 22323303
- [Background] O'Brien LM, Mervis CB, Holbrook CR, Bruner JL, Smith NH, McNally N, McClimment MC, Gozal D. Neurobehavioral correlates of sleep-disordered breathing in children. J Sleep Res. 2004 Jun;13(2):165-72. doi: 10.1111/j.1365-2869.2004.00395.x. PMID 15175097
- [Background] Gozal D. Sleep-disordered breathing and school performance in children. Pediatrics. 1998 Sep;102(3 Pt 1):616-20. doi: 10.1542/peds.102.3.616. PMID 9738185
- [Background] Marcus CL, Moore RH, Rosen CL, Giordani B, Garetz SL, Taylor HG, Mitchell RB, Amin R, Katz ES, Arens R, Paruthi S, Muzumdar H, Gozal D, Thomas NH, Ware J, Beebe D, Snyder K, Elden L, Sprecher RC, Willging P, Jones D, Bent JP, Hoban T, Chervin RD, Ellenberg SS, Redline S; Childhood Adenotonsillectomy Trial (CHAT). A randomized trial of adenotonsillectomy for childhood sleep apnea. N Engl J Med. 2013 Jun 20;368(25):2366-76. doi: 10.1056/NEJMoa1215881. Epub 2013 May 21. PMID 23692173
- [Background] Glasson EJ, Jacques A, Wong K, Bourke J, Leonard H. Improved Survival in Down Syndrome over the Last 60 Years and the Impact of Perinatal Factors in Recent Decades. J Pediatr. 2016 Feb;169:214-20.e1. doi: 10.1016/j.jpeds.2015.10.083. Epub 2015 Dec 2. PMID 26651430
- [Background] Kucik JE, Shin M, Siffel C, Marengo L, Correa A; Congenital Anomaly Multistate Prevalence and Survival Collaborative. Trends in survival among children with Down syndrome in 10 regions of the United States. Pediatrics. 2013 Jan;131(1):e27-36. doi: 10.1542/peds.2012-1616. Epub 2012 Dec 17. PMID 23248222
- [Background] Rajagopal KR, Abbrecht PH, Derderian SS, Pickett C, Hofeldt F, Tellis CJ, Zwillich CW. Obstructive sleep apnea in hypothyroidism. Ann Intern Med. 1984 Oct;101(4):491-4. doi: 10.7326/0003-4819-101-4-491. PMID 6476635
- [Background] Stebbens VA, Dennis J, Samuels MP, Croft CB, Southall DP. Sleep related upper airway obstruction in a cohort with Down's syndrome. Arch Dis Child. 1991 Nov;66(11):1333-8. doi: 10.1136/adc.66.11.1333. PMID 1836718
- [Background] Marcus CL, Keens TG, Bautista DB, von Pechmann WS, Ward SL. Obstructive sleep apnea in children with Down syndrome. Pediatrics. 1991 Jul;88(1):132-9. PMID 1829151
- [Background] de Miguel-Diez J, Villa-Asensi JR, Alvarez-Sala JL. Prevalence of sleep-disordered breathing in children with Down syndrome: polygraphic findings in 108 children. Sleep. 2003 Dec 15;26(8):1006-9. doi: 10.1093/sleep/26.8.1006. PMID 14746382
- [Background] Redline S, Tishler PV, Schluchter M, Aylor J, Clark K, Graham G. Risk factors for sleep-disordered breathing in children. Associations with obesity, race, and respiratory problems. Am J Respir Crit Care Med. 1999 May;159(5 Pt 1):1527-32. doi: 10.1164/ajrccm.159.5.9809079. PMID 10228121
- [Background] Marcus CL, Brooks LJ, Draper KA, Gozal D, Halbower AC, Jones J, Schechter MS, Ward SD, Sheldon SH, Shiffman RN, Lehmann C, Spruyt K; American Academy of Pediatrics. Diagnosis and management of childhood obstructive sleep apnea syndrome. Pediatrics. 2012 Sep;130(3):e714-55. doi: 10.1542/peds.2012-1672. Epub 2012 Aug 27. PMID 22926176
- [Background] Farhood Z, Isley JW, Ong AA, Nguyen SA, Camilon TJ, LaRosa AC, White DR. Adenotonsillectomy outcomes in patients with Down syndrome and obstructive sleep apnea. Laryngoscope. 2017 Jun;127(6):1465-1470. doi: 10.1002/lary.26398. Epub 2017 Jan 5. PMID 28055122
- [Background] Hawkins SM, Jensen EL, Simon SL, Friedman NR. Correlates of Pediatric CPAP Adherence. J Clin Sleep Med. 2016 Jun 15;12(6):879-84. doi: 10.5664/jcsm.5892. PMID 27092702
- [Background] Marcus CL, Brooks LJ, Draper KA, Gozal D, Halbower AC, Jones J, Schechter MS, Sheldon SH, Spruyt K, Ward SD, Lehmann C, Shiffman RN; American Academy of Pediatrics. Diagnosis and management of childhood obstructive sleep apnea syndrome. Pediatrics. 2012 Sep;130(3):576-84. doi: 10.1542/peds.2012-1671. Epub 2012 Aug 27. PMID 22926173
- [Background] Marcus CL, Beck SE, Traylor J, Cornaglia MA, Meltzer LJ, DiFeo N, Karamessinis LR, Samuel J, Falvo J, DiMaria M, Gallagher PR, Beris H, Menello MK. Randomized, double-blind clinical trial of two different modes of positive airway pressure therapy on adherence and efficacy in children. J Clin Sleep Med. 2012 Feb 15;8(1):37-42. doi: 10.5664/jcsm.1656. PMID 22334807
- [Background] Strydom A, Coppus A, Blesa R, Danek A, Fortea J, Hardy J, Levin J, Nuebling G, Rebillat AS, Ritchie C, van Duijn C, Zaman S, Zetterberg H. Alzheimer's disease in Down syndrome: An overlooked population for prevention trials. Alzheimers Dement (N Y). 2018 Dec 13;4:703-713. doi: 10.1016/j.trci.2018.10.006. eCollection 2018. PMID 30581976
- [Background] Sawyer AM, Gooneratne NS, Marcus CL, Ofer D, Richards KC, Weaver TE. A systematic review of CPAP adherence across age groups: clinical and empiric insights for developing CPAP adherence interventions. Sleep Med Rev. 2011 Dec;15(6):343-56. doi: 10.1016/j.smrv.2011.01.003. Epub 2011 Jun 8. PMID 21652236
- [Background] O'Donnell AR, Bjornson CL, Bohn SG, Kirk VG. Compliance rates in children using noninvasive continuous positive airway pressure. Sleep. 2006 May;29(5):651-8. PMID 16774155
- [Background] Castro-Codesal ML, Dehaan K, Featherstone R, Bedi PK, Martinez Carrasco C, Katz SL, Chan EY, Bendiak GN, Almeida FR, Olmstead DL, Young R, Woolf V, Waters KA, Sullivan C, Hartling L, MacLean JE. Long-term non-invasive ventilation therapies in children: A scoping review. Sleep Med Rev. 2018 Feb;37:148-158. doi: 10.1016/j.smrv.2017.02.005. Epub 2017 Mar 2. PMID 28410811
- [Background] Nixon GM, Mihai R, Verginis N, Davey MJ. Patterns of continuous positive airway pressure adherence during the first 3 months of treatment in children. J Pediatr. 2011 Nov;159(5):802-7. doi: 10.1016/j.jpeds.2011.04.013. Epub 2011 May 20. PMID 21601219
- [Background] Marcus CL, Ward SL, Mallory GB, Rosen CL, Beckerman RC, Weese-Mayer DE, Brouillette RT, Trang HT, Brooks LJ. Use of nasal continuous positive airway pressure as treatment of childhood obstructive sleep apnea. J Pediatr. 1995 Jul;127(1):88-94. doi: 10.1016/s0022-3476(95)70262-8. PMID 7608817
- [Background] Kang EK, Xanthopoulos MS, Kim JY, Arevalo C, Shults J, Beck SE, Marcus CL, Tapia IE. Adherence to Positive Airway Pressure for the Treatment of Obstructive Sleep Apnea in Children With Developmental Disabilities. J Clin Sleep Med. 2019 Jun 15;15(6):915-921. doi: 10.5664/jcsm.7850. PMID 31138379
- [Background] Boeije H. A purposeful approach to the constant comparative method in the analysis of qualitative interviews. Quality and Quantity. 2002;36:391-409
- [Derived] Xanthopoulos MS, Nelson MN, Eriksen W, Barg FK, Byars KC, Ishman SL, Esbensen AJ, Meinzen-Derr J, Heubi CH, Gurbani NS, Bradford R, Hicks S, Tapia IE. Caregiver experiences helping children with Down syndrome use positive airway pressure to treat obstructive sleep apnea. Sleep Med. 2023 Jul;107:179-186. doi: 10.1016/j.sleep.2023.04.022. Epub 2023 Apr 28. PMID 37196396

RESULTS

PARTICIPANT FLOW:
Groups:
- Interview Completion: The number of participants who completed the interview process.
Period: Overall Study
Arm/Group | Interview Completion
Started | 42
Completed | 41
Not Completed | 1
Not completed — screen failure | 1

BASELINE CHARACTERISTICS:
Population: The number of participants who completed the interview process from both study sites.
Arm/Group | Interview Completion
Number analyzed (Participants) | 41
Age, Customized [Mean (Standard Deviation); unit: years]
  Age at screening | 12.6 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  All Sites: Female | 28
  All Sites: Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  All Sites: Hispanic or Latino | 0
  All Sites: Not Hispanic or Latino | 41
  All Sites: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  All Sites: American Indian or Alaska Native | 0
  All Sites: Asian | 2
  All Sites: Native Hawaiian or Other Pacific Islander | 0
  All Sites: Black or African American | 10
  All Sites: White | 29
  All Sites: More than one race | 0
  All Sites: Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed Interviews Regarding Positive Airway Pressure (PAP) Acceptability
Description: PAP feasibility will be measured by completion of semi-structured interviews to explore attitudes about PAP therapy in youth with Down Syndrome and Obstructive Sleep Apnea Syndrome.
Time Frame: one day
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Completion
Number analyzed (Participants) | 41
Participants
  Site 1 -- CHOP | 20
  Site 2 -- Cincinnati Children's Hospital | 21

ADVERSE EVENTS:
Time Frame: Up to one hour
Description: There were no adverse events reported as this is a one-time telephone interview study.
Arm/Group | Interview Completion
All-Cause Mortality (participants affected / at risk) | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT04124471/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT04124471/ICF_001.pdf